CLINICAL TRIAL: NCT00004249
Title: Immunization Using Polysialic Acid-KLH or N-Propionylated Polysialic Acid-KLH Conjugate Plus the Immunological Adjuvant QS-21 in Patients With Small Cell Lung Cancer Who Have Achieved a Major Response to Initial Therapy
Brief Title: Vaccine Therapy Plus QS21 in Treating Patients With Small Cell Lung Cancer That Has Responded to Initial Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 98-065; CDR0000067495 (Registry Identifier: PDQ (Physician Data Query)); NCI-H99-0047
Record Dates: First submitted 2000-01-28; First posted 2004-04-28 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — saponin QA-21V1; keyhole-limpet hemocyanin; polysialic acid

INTERVENTIONS:
Biological: QS21
Biological: keyhole limpet hemocyanin
Drug: polysialic acid

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Biological therapies, such as QS21, use different ways to stimulate the immune system and stop cancer cells from growing.

PURPOSE: Phase II trial to study the effectiveness of vaccine therapy plus QS21 in treating patients who have small cell lung cancer that has responded to initial therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the antibody response after immunization with polysialic acid keyhole limpet hemocyanin (PSA-KLH) conjugate or N-propionylated PSA-KLH conjugate plus immunological adjuvant QS21 in patients with small cell lung cancer. II. Assess the clinical toxicities resulting from these regimens and from the immune response in this patient population.

OUTLINE: Patients receive polysialic acid keyhole limpet hemocyanin (PSA-KLH) conjugate or N-propionylated PSA-KLH conjugate plus immunological adjuvant QS21 subcutaneously weekly on weeks 1-4 and on weeks 8 and 16 for a total of 6 vaccinations. Patients are followed at 2 weeks, and then every 3 months for up to 1 year.

PROJECTED ACCRUAL: A total of 12 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed small cell lung cancer Must have completed initial therapy with or without radiotherapy and have achieved a complete response or partial response to therapy without subsequent evidence of disease progression Must have completed any radiotherapy including prophylactic cranial radiotherapy as part of the planned primary therapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Lymphocyte count at least 500/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT no greater than 1.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 1.5 times ULN Renal: Not specified Cardiovascular: No New York Heart Association class III or IV heart disease Other: No known immunodeficiency or autoimmune disease No other active malignancies within the past 5 years except nonmelanoma skin cancer No clinically significant peripheral neuropathy Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics At least 4 weeks but no more than 12 weeks since prior initial therapy and recovered Chemotherapy: See Disease Characteristics At least 4 weeks but no more than 12 weeks since prior initial therapy and recovered Endocrine therapy: See Disease Characteristics At least 4 weeks but no more than 12 weeks since prior initial therapy and recovered No concurrent corticosteroids Radiotherapy: See Disease Characteristics At least 4 weeks but no more than 12 weeks since prior initial therapy and recovered No prior radiotherapy to the spleen Surgery: No prior splenectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-08; Primary Completion 2001-11 (Actual); Study Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee M. Krug, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States